### **Informed Consent Form (ICF)**

Study Title: Comparison of Postoperative Pulmonary Complications Between Smokers and Nonsmokers: A

**Prospective Cohort Study** 

NCT Number: NCT06982911

Date: May 2025

# INFORMATION FOR PARTICIPANTS

You are invited to participate in a research study. Your participation is entirely voluntary. Before you decide whether or not to participate, please take time to read the following information carefully. It explains the purpose of the study, how your data will be used, what the study involves, and any potential benefits or risks. If you agree to participate, please sign the informed consent section at the end. You are free to withdraw from the study at any time. No payment will be made to you, and you will not be expected to provide any financial or material contribution.

### PURPOSE OF THE STUDY

This study aims to investigate the role of smoking in the development of postoperative pulmonary complications (PPCs). A total of 70 patients undergoing surgery at Gazi Yasargil Training and Research Hospital will be included. The estimated observation period per participant is approximately 3 hours.

### **STUDY PROCEDURES**

This is an observational study. No intervention or procedure will be performed outside of standard routine clinical care.

#### **POTENTIAL BENEFITS**

Participants in this study will contribute to the understanding of the impact of smoking on postoperative outcomes. However, there may be no direct benefit to you.

#### **COST OF PARTICIPATION**

Participation in this study will not result in any financial burden. No payment will be provided.

## **VOLUNTARY PARTICIPATION**

Your participation is completely voluntary. Even if you sign this form now, you may withdraw from the study at any time without providing a reason. If you decide not to participate or to withdraw later, your medical care and treatment will not be affected. Similarly, the investigator may withdraw you from the study if it is deemed not in your best interest.

#### **CONFIDENTIALITY**

Your personal information will be kept confidential and used only for the purposes of research and statistical analysis. Only the study team will have access to this data, unless it is required by an ethics committee or legal authority. The results of the study may be published in medical literature, but your identity will not be revealed. You also have the right to access your own study-related data.

#### **OUESTIONS OR CONCERNS**

Contact Person:

Name: Dr. Mehmet Özkılıç

Title: Specialist in Anesthesiology and Reanimation

Phone: +90 507 006 83 13

### PARTICIPANT CONSENT

I have discussed this study in detail with the investigator and had all my questions answered. I have read and understood this informed consent form. I voluntarily agree to participate in this study and sign this form of my own free will. I understand that signing this form does not waive any of my legal rights. I have received a copy of this form for my own reference.

| Participant Name: |
|---------------------------------|
| Date and Signature: |
| Phone: |
| Legal Guardian (if applicable): |
| Date and Signature: |
| Phone: |

Witness Name:

| Data | a | Cian | 041110 |
|------|-----|-------|--------|
| Date | anu | 21511 | ature: |

Phone:

Investigator Name: Dr. Mehmet Özkılıç

Date and Signature:

Phone: +90 507 006 83 13

\*Note:\* The witness is the person who observed the informed consent process from start to finish. The investigator is the person who informed the participant about the study.